CLINICAL TRIAL: NCT04157946
Title: Risk Assessment of Ventilator-induced Lung Injury in Patients With Acute Respiratory Distress Syndrome: The Role of Morphological Phenotype in ARDS
Brief Title: The Role of Morphological Phenotype in ARDS
Acronym: MPARDS
Status: Completed | Type: Observational
Sponsor: Hospital El Cruce (Other)
Responsible Party: Principal Investigator, Nestor Pistillo, Head of Intensive Care Unit at Hospital El Cruce, Hospital El Cruce
Other Study IDs: HElCruce
Record Dates: First submitted 2019-11-05; First posted 2019-11-08 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-11

CONDITIONS: Respiratory Distress Syndrome, Adult
Keywords: Respiratory Insufficiency; Ventilator-Induced Lung Injury; Ventilators, Mechanical
MeSH Terms: conditions — Respiratory Distress Syndrome; Respiratory Insufficiency; Ventilator-Induced Lung Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Focal: ARDS was classified according to the pattern that adopted the loss of aeration in the chest CT in the two groups: focal (predominant commitment in the dependant region) and non- focal (patched or diffused involvement of the entire lung)
  Interventions: Diagnostic Test: CT
- Non-Focal: ARDS was classified according to the pattern that adopted the loss of aeration in the chest CT in the two groups: focal (predominant commitment in the dependant region) and non- focal (patched or diffused involvement of the entire lung)
  Interventions: Diagnostic Test: CT

INTERVENTIONS:
Diagnostic Test: CT — Patients with ARDS were included. We excluded patients with emphysema, asthma, pneumothorax, or serious conditions of instability: oxygen saturation ≤ 88%; severe shock, ventricular arrhythmia, or myocardial ischemia.
  To allow comparison between groups, patients were ventilated in volume control under similar conditions of tidal volume (TV; 6 ml/kg-PBW), plateau pressure (PPlat 30 cmH2O), respiratory rate (18 bit/min) and constant flow. PEEP was adjusted to reach objective PPlat.
  Transpulmonary pressures (TP) were measured and a chest CT scan performed during an expiratory and inspiratory pause. Global and regional volumes of lungs were measured using specific software (Volume Analysis Software,Toshiba, Japan). Three regions were identified: basal (from the diaphragm to the carina), middle (from the carina to the aortic arch) and apical (above the aortic arch).
  Other Names: Transpulmonary pressures (TP) were measured

SUMMARY:
Although most of the information focuses on understanding how the ventilator produces lung damage, the pulmonary factors that predispose to ventilator-induced lung injury (VILI) have been less studied. Acute respiratory distress syndrome (ARDS) can adopt different morphological phenotypes, with its own clinical and mechanical characteristics. This morphological phenotypes may favor the development of VILI for same ventilatory strategy

DETAILED DESCRIPTION:
The lung in acute respiratory distress syndrome ARDS) is a heterogeneous viscoelastic system, in which areas with different time constants coexist, causing tidal volume to be distributed unevenly within an anatomically and functionally reduced lung. The administration of a disproportionately high tidal volume for this lung predisposes to the over-distension of the better ventilated alveoli and to the injury by tidal opening and closing of the alveoli more unstable. In this sense, using low tidal volume and homogenizing the lung by means of the prone position have proven beneficial in ARDS.

Tidal volume, driving pressure, inspiratory flow and respiratory rate have been identified as responsible for mechanical ventilation-induced lung injury (VILI). These factors together represent the mechanical power, the insulting energy which is repeatedly applied to a vulnerable lung parenchyma.

Although most of the information focuses on understanding how the ventilator produces lung damage and/or amplifies the existing one, the pulmonary factors that predispose to VILI have been less studied. Acute respiratory distress syndrome can adopt different morphological phenotypes, with its own clinical and mechanical characteristics. Understanding how each subgroup of ARDS responds to the protective ventilatory strategy could help to personalize treatment.

Objectives: To compare the risk of VILI in two groups of ARDS with different morphological phenotypes (focal and non-focal), ventilated with the same protective strategy.

Design: Patients with ARDS were ventilated under the same conditions of both tidal volume (TV) and plateau pressure (PPlat). Positive End Expiratory Pressure (PEEP) was adjusted to reach 30 cmH2O of PPlat. A CT was performed in inspiration and expiration. Transpulmonary pressures (TP) were measured and lung volumes calculated (Volume Analysis Software,Toshiba, Japan). Stress was defined as TP at the end of inspiration (TPinsp) and strain: tidal volume/End Expiratory Lung Volume Patients were classified into focal and non-focal according to the distribution of aeration loss in CT. Mann - Whitney U test was used to compare variables and Pearson correlation coefficient to compare its correlation. Significant: p <0.05

ELIGIBILITY:
Inclusion Criteria:

Acute respiratory distress syndrome (ARDS).

Exclusion Criteria:

Emphysema Asthma Pneumothorax Oxygen saturation ≤ 88% Severe shock Ventricular arrhythmia Myocardial ischemia.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with moderate to severe ARDS diagnosis were studied according to the Berlin definition. The AECC defined ARDS as the acute onset of hypoxemia (arterial partial pressure of oxygen to fraction of inspired oxygen [PaO2/FIO2] ≤ 200 mm Hg) with bilateral infiltrates on frontal chest radiograph, with no evidence of left atrial hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2017-08-07 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-20 (Actual)

PRIMARY OUTCOMES:
Measuring the level of pulmonary stress caused by mechanical ventilation | One year
  Twelve patients with ARDS were studied (six from each group). A balloon catheter was placed at the distal end of the esophagus to measure esophageal pressures. A pneumotachograph was used to record and quantify esophageal pressures during the ventilatory cycle. Esophageal pressure is considered as equivalent of pleural pressure. Pulmonary distention pressure (transpulmonary pressure) is obtained by measuring the difference between the pressure of the respiratory system (supplied by mechanical ventilation) and esophageal pressure. Stress was defined as the transpulmonary pressure measure at the end of an inspiratory pause (in zero flow conditions). Pulmonary stress was quantified in cmH2O. There is a linear relationship between stress and lung damage (VILI). Mann-Whitney U test was used to compare variables. Significant p < 0.05.
Measurement of pulmonary strain caused by mechanical ventilation | One year
  Twelve patients with ARDS were studied (six from each group). A chest tomography was performed during an expiratory and inspiratory pause. Using a specific software (Lung Volume Analysis Software.Toshiba, Japan), the amount of lung volume was calculated in expiration and inspiration air (expressed in ml). The strain was defined as the relationship between the amount of volume supplied by mechanical ventilation (tidal volume) and the lung's ability to receive that volume (EELV: end expiratory lung volume). This ratio was expressed as a percentage. There is a direct relationship between strain and lung damage (VILI). Mann-Whitney U test was used to compare variables. Significant p < 0.05..
Measurement of injury due to cyclic opening and closing of the most unstable caused by mechanical ventilation . | One year
  Twelve patients with ARDS were studied (six from each group). Three lung regions were studied on tomography: Basal, middle and apical. A specific software quantified the amount of airless lung (100 to - 100 HU), both in expiration and inspiration. This amount was expressed in numbers of pixels. A lesion due to cyclic opening and closing of the alveoli was defined as the difference between the size of the airless lung between both respiratory times, in relation to the basal condition (lung without air at expiration). This ratio was expressed as a percentage. There is a direct relationship between this mechanism of damage and the risk of VILI. Mann-Whitney U test was used to compare variables. Significant p < 0.05.

SECONDARY OUTCOMES:
Measurement of pulmonary hyperinflation caused by mechanical ventilation | One year
  Twelve patients with ARDS were studied (six from each group). Lung regions were studied on tomography: Basal, middle and apical. A specific software was quantified the amount of excess air (hyperinflation:-900 to - 1000 HU). Hyperinflation was expressed in relation to the total lung volume as a percentage. There is a direct relationship between hyperinflation and the risk of VILI. Mann-Whitney U test was used to compare variables. Significant p < 0.05.

CONTACTS AND LOCATIONS:
Overall Officials: Nestor Pistillo, MD, Principal Investigator — Hospital El Cruce
Locations (1):
- Hospital El Cruce, San Juan Bautista, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guerin C, Beuret P, Constantin JM, Bellani G, Garcia-Olivares P, Roca O, Meertens JH, Maia PA, Becher T, Peterson J, Larsson A, Gurjar M, Hajjej Z, Kovari F, Assiri AH, Mainas E, Hasan MS, Morocho-Tutillo DR, Baboi L, Chretien JM, Francois G, Ayzac L, Chen L, Brochard L, Mercat A; investigators of the APRONET Study Group, the REVA Network, the Reseau recherche de la Societe Francaise d'Anesthesie-Reanimation (SFAR-recherche) and the ESICM Trials Group. A prospective international observational prevalence study on prone positioning of ARDS patients: the APRONET (ARDS Prone Position Network) study. Intensive Care Med. 2018 Jan;44(1):22-37. doi: 10.1007/s00134-017-4996-5. Epub 2017 Dec 7. PMID 29218379
- [Background] Protti A, Andreis DT, Monti M, Santini A, Sparacino CC, Langer T, Votta E, Gatti S, Lombardi L, Leopardi O, Masson S, Cressoni M, Gattinoni L. Lung stress and strain during mechanical ventilation: any difference between statics and dynamics? Crit Care Med. 2013 Apr;41(4):1046-55. doi: 10.1097/CCM.0b013e31827417a6. PMID 23385096
- [Background] Cressoni M, Cadringher P, Chiurazzi C, Amini M, Gallazzi E, Marino A, Brioni M, Carlesso E, Chiumello D, Quintel M, Bugedo G, Gattinoni L. Lung inhomogeneity in patients with acute respiratory distress syndrome. Am J Respir Crit Care Med. 2014 Jan 15;189(2):149-58. doi: 10.1164/rccm.201308-1567OC. PMID 24261322
- [Background] Gattinoni L, Marini JJ, Pesenti A, Quintel M, Mancebo J, Brochard L. The "baby lung" became an adult. Intensive Care Med. 2016 May;42(5):663-673. doi: 10.1007/s00134-015-4200-8. Epub 2016 Jan 18. PMID 26781952
- [Background] Acute Respiratory Distress Syndrome Network; Brower RG, Matthay MA, Morris A, Schoenfeld D, Thompson BT, Wheeler A. Ventilation with lower tidal volumes as compared with traditional tidal volumes for acute lung injury and the acute respiratory distress syndrome. N Engl J Med. 2000 May 4;342(18):1301-8. doi: 10.1056/NEJM200005043421801. PMID 10793162
- [Background] Nieman GF, Satalin J, Andrews P, Habashi NM, Gatto LA. Lung stress, strain, and energy load: engineering concepts to understand the mechanism of ventilator-induced lung injury (VILI). Intensive Care Med Exp. 2016 Dec;4(1):16. doi: 10.1186/s40635-016-0090-5. Epub 2016 Jun 18. PMID 27316442
- [Background] Retamal J, Hurtado D, Villarroel N, Bruhn A, Bugedo G, Amato MBP, Costa ELV, Hedenstierna G, Larsson A, Borges JB. Does Regional Lung Strain Correlate With Regional Inflammation in Acute Respiratory Distress Syndrome During Nonprotective Ventilation? An Experimental Porcine Study. Crit Care Med. 2018 Jun;46(6):e591-e599. doi: 10.1097/CCM.0000000000003072. PMID 29528946
- [Result] ARDS Definition Task Force; Ranieri VM, Rubenfeld GD, Thompson BT, Ferguson ND, Caldwell E, Fan E, Camporota L, Slutsky AS. Acute respiratory distress syndrome: the Berlin Definition. JAMA. 2012 Jun 20;307(23):2526-33. doi: 10.1001/jama.2012.5669. PMID 22797452